CLINICAL TRIAL: NCT06207045
Title: The Effects of Limb Elevation During Gout Flare Episodes : A Pilot, Randomised Controlled Trial
Brief Title: The Effects of Limb Elevation During Gout Flare Episodes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, saitip sangkamanovet, Dr., Thammasat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTU-EC-IM-4-290/66
Record Dates: First submitted 2024-01-05; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Gout Flare
Keywords: Gout, arthritis, gout flare
MeSH Terms: conditions — Gout; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- limb elevation group (Experimental): limb elevation plus standard medication
  Interventions: Procedure: limb elevation
- control group (No Intervention): standard medication only

INTERVENTIONS:
Procedure: limb elevation — limb elevation more than 45 degrees
  Arms: limb elevation group

SUMMARY:
The goal of this open-label randomized controlled trial is to explore the benefit of limb elevation in inpatient gout flare episodes, compared with standard treatment The main questions are;

* Is limb elevation able to reduce pain during gout flare episodes to a greater degree compared with standard treatment ?
* Is Is limb elevation able to reduce joint swelling during gout flare episodes to a greater degree compared with standard treatment ?

Participants will be divided into 2 group;

1. Limb elevation group
2. control group All participants will receive standard medical therapy consisting of colchicine 0.6 mg per day plus prednisolone 30 mg per day for 2 days

Pain score and joint circumference will be recored at recruitment, 24 hour and 48 hour

DETAILED DESCRIPTION:
Limb elevation has shown benefit in ankle sprain and venous insufficiency, but its benefit has not been studied in people with gout flare. In this open-label randomized controlled trial, 30 adults diagnosed with gout flare during their hospitalization will be randomized to receive limb elevation plus standard medication for gout flare (limb elevation group) or standard medication only (control group). Primary outcome is reduction in 10-point visual analogue scale for pain at 48 hours after enrollment and the secondary outcome is the reduction of the circumference of affected joint at 48 hours after enrollment. Comparison of pain score and joint circumference reduction will be made using Wilcoxon Rank-sum test. Our study results may provide some evidence in support of limb elevation as a supplementary non-pharmacological therapy for relief of gout flare.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Diagnosis of Gout according to 2015 The ACR/EULAR gout classification criteria

Exclusion Criteria:

* Receive Non-Steroidal Anti-inflammatory Drugs or Intra-articular corticosteroids or prednisolone > 10 mg within 24 hours before enrollment
* Unstable vital sign
* Receiving joint aspiration for release joint effusion ≥ 10 ml after enrollment
* Gout flares involve axial joints e.g. hip
* Glomerular Filtration Rates < 30 ml/min/1.73m2
* Communication problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain score | 48 hours
  10-points Visual Analogue Scale

SECONDARY OUTCOMES:
Joint circumference | 48 hours
  circumference of affected joint in centimeter

CONTACTS AND LOCATIONS:
Overall Officials: saitip sangkamanovet, Principal Investigator — Thammasat University
Locations (1):
- Thammasat University, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No